CLINICAL TRIAL: NCT07050381
Title: Risk Factors Related to Rupture Flow-related Aneurysms in Posterior Arteriovenious Malformation: A Muti-center Observentional Research.
Brief Title: The Risk Factors Related to Rupture Flow-related Aneurysms in Posterior AVM
Acronym: pAVM-rFA
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Lu Hua, professor, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: pAVM-rFA
Record Dates: First submitted 2025-02-10; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Arteriovenous Malformation of Central Nervous System; Aneurysm, Ruptured; Aneurysmatic Subarachnoid Haemorrhage; Aneurysm Cerebral
Keywords: arteriovenous malformation; flow-related aneurysm; ruptured aneurysm; subarachnoid hemorrhage
MeSH Terms: conditions — Aneurysm, Ruptured; Intracranial Aneurysm; Arteriovenous Malformations; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- pAVM with ruptured flow-related aneurysm
- pAVM without ruptured flow-related aneurysm

SUMMARY:
AVMs have been reported to rupture at a formidable annual rate of 2% to 3% at natural progression, often resulting in longterm neurological deficits and poor functional outcomes.The reported risk of hemorrhagic presentation in patients with AVMs is 41% to 65%. While many studies suggest a correlation between higher hemorrhage risk and the concurrent presence of AVM and aneurysms, few authors have focused specifically on flow-related aneurysms alone. In many instances, the source of rupture is also unclear. Meta-analysis from 2016 suggested that 49.2% of hemorrhages were secondary to aneurysm rupture, 45% from AVM rupture, and 5.7% were undetermined.In a study of 302 patients, of which 52.6% had a hemorrhagic presentation, demonstrated a significant increase in rate of hemorrhage in those with flow-related aneurysms. Thus, it is necessary to figure out risk factors related to ruptured flow-related aneurysms in pAVM.

ELIGIBILITY:
Inclusion Criteria:

1. pAVM with flow-related aneurysms were identified by DSA, and subarachnoid hemorrhage was confirmed by CT
2. No history of stroke, Marfan syndrome, polycystic kidney disease

Exclusion Criteria:

1. pAVM without flow-related aneurysms
2. Absence of clinical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with posterior circulation malformations combined with ruptured or unruptured flow-related aneurysms will be included. Morphological data such as aneurysm size, location, parent artery, feeding arteries, draining vein count, malformation size, malformation location, and the ratio of malformation/aneurysm volume will be analyzed. These factors will be examined alongside medical histories of hypertension, diabetes, and coronary artery disease to investigate the risk factors for ruptured flow-related aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
characteristics of flow-related aneurysm | From enrollment to the end of treatment at 8 weeks
  size ratio(aneurysm depth (mm)/parent artery diameter (mm))

OTHER OUTCOMES:
demographic information of pAVM-rFA | From enrollment to the end of treatment at 8 weeks
  gender
demographic information | From enrollment to the end of treatment at 8 weeks
  age when be hospitalized
characteristics of flow-related aneurysm | From enrollment to the end of treatment at 8 weeks
  aspect ratio (aneurysm depth (mm)/aneurysm neck (mm))
characteristic of avm | From enrollment to the end of treatment at 8 weeks
  avm location
characteristic of avm | From enrollment to the end of treatment at 8 weeks
  Spetzler-Martin grade of avm

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hung AL, Yang W, Jiang B, Garzon-Muvdi T, Caplan JM, Colby GP, Coon AL, Tamargo RJ, Huang J. The Effect of Flow-Related Aneurysms on Hemorrhagic Risk of Intracranial Arteriovenous Malformations. Neurosurgery. 2019 Oct 1;85(4):466-475. doi: 10.1093/neuros/nyy360. PMID 30107479
- [Background] Shakur SF, Amin-Hanjani S, Mostafa H, Charbel FT, Alaraj A. Hemodynamic Characteristics of Cerebral Arteriovenous Malformation Feeder Vessels With and Without Aneurysms. Stroke. 2015 Jul;46(7):1997-9. doi: 10.1161/STROKEAHA.115.009545. Epub 2015 May 19. PMID 25991417
- [Background] Kouznetsov E, Weill A, Ghostine JS, Gentric JC, Raymond J, Roy D. Association between posterior fossa arteriovenous malformations and prenidal aneurysm rupture: potential impact on management. Neurosurg Focus. 2014 Sep;37(3):E4. doi: 10.3171/2014.6.FOCUS14219. PMID 25175442
- [Background] Lv X, Wu Z, Jiang C, Yang X, Li Y, Sun Y, Zhang N. Angioarchitectural characteristics of brain arteriovenous malformations with and without hemorrhage. World Neurosurg. 2011 Jul-Aug;76(1-2):95-9. doi: 10.1016/j.wneu.2011.01.044. PMID 21839959